CLINICAL TRIAL: NCT05009641
Title: Carnitine Supplementation and Skeletal Muscle Function in Aging
Brief Title: Carnitine Supplementation and Skeletal Muscle Mass
Acronym: ROM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gdansk University of Physical Education and Sport (Other)
Collaborators: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Robert Olek, Principal Investigator, Gdansk University of Physical Education and Sport
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCN_ROM; 2014/15/B/NZ7/00893 (Other Grant/Funding Number: National Science Centre)
Record Dates: First submitted 2021-08-05; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Muscle Loss
MeSH Terms: conditions — Muscular Atrophy | interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- carnitine2 (Experimental): 2000 mg L-carnitine per day for 24 weeks
  Interventions: Dietary Supplement: L-carnitine
- carnitine (Active Comparator): 1000 mg L-carnitine per day for 24 weeks
  Interventions: Dietary Supplement: L-carnitine
- control (No Intervention): no supplementation

INTERVENTIONS:
Dietary Supplement: L-carnitine
  Other Names: L-carnitine-L-tartrate
  Arms: carnitine; carnitine2

SUMMARY:
The primary aim of the current research project is to investigate the effect of carnitine supplementation on muscle strength and body composition.

A secondary aim of this project is to explore the effect of circulating trimethylamine N-oxide elevation, induced by carnitine supplementation on muscle strength and body composition.

ELIGIBILITY:
Inclusion Criteria:

* must be able to swallow tablets

Exclusion Criteria:

* cardiovascular disease
* liver disease
* kidney disease
* neuromuscular disease
* gastrointestinal disorders (including stomach ulcers and erosions)
* diabetes
* other severe chronic diseases

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-11-15 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Muscle Strength using Biodex System 4 Pro dynamometer | 24 weeks
  Peak torque measured by performing maximum voluntary contractions during isometric knee extension and flexion. The test performed in concentric-concentric mode consisting maximum 4-s knee extensor isometric contraction and maximum 4-s knee flexor isometric contraction, separated by 20-s recovery, repeated three times. Muscle isokinetic strength assessed in 5 repetitions of flexion and extension at a speed of 60°/s. Muscle endurance assessed in 10 repetitions at 300°/s determine the ability of the muscle to maintain the work. Strength testing performed on the Biodex System 4 Pro dynamometer.
Body Composition: Body Fat Mass, Fat Free Mass, and Skeletal Muscle Mass using a bioelectrical impedance analyzer (InBody720) | 24 weeks
  The InBody720 measures impedance of five segments of the body (each arm, each leg, trunk) at frequencies of 1, 5, 50, 250, 500, and 1000 kHz through the 8-polar tactile-electrode. Based on the impedance, body fat mass, fat free mass, and skeletal muscle mass are calculated.

SECONDARY OUTCOMES:
Plasma trimethylamine N-oxide concentration | 24 weeks
  Blood samples taken before the start and after finishing the supplementation protocol. Plasma trimethylamine N-oxide determined using ultra performance liquid chromatography - tandem mass spectrometer (UPLC-MS/MS) method